CLINICAL TRIAL: NCT01430741
Title: MISSION-Vet HUD-VASH Implementation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SDP 11-240
Record Dates: First submitted 2011-07-26; First posted 2011-09-08 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-05

CONDITIONS: Substance Related Disorders; Mental Illness
Keywords: Implementation Science; Supportive Housing; Co-occurring disorders; Cluster randomized controlled trial; Hybrid implementation-effectiveness trial
MeSH Terms: conditions — Substance-Related Disorders; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Implementation as Usual Case Management (Other): Maintaining Independence and Sobriety Through Systems Integration, Outreach, and Networking (Veterans Edition):MISSION-Vet has been developed to target mental health, substance abuse and related issues faced by homeless Veterans through assertive outreach, psychoeducation, and linkages to community-based resources.
  Implementation as Usual (IU) - standard training on the MISSION model via a 1.5 hour webinar
  Interventions: Behavioral: Maintaining Independence and Sobriety Through Systems Integration, Outreach, and Networking (Veterans Edition)
- Implementation as Usual Veterans (Other): Maintaining Independence and Sobriety Through Systems Integration, Outreach, and Networking (Veterans Edition):MISSION-Vet has been developed to target mental health, substance abuse and related issues faced by homeless Veterans through assertive outreach, psychoeducation, and linkages to community-based resources.
  Implementation as Usual (IU) - standard training on the MISSION model via a 1.5 hour webinar. Staff then deliver MISSION to Veterans.
  Interventions: Behavioral: Maintaining Independence and Sobriety Through Systems Integration, Outreach, and Networking (Veterans Edition)
- Getting to Outcomes Case Management (Experimental): Getting To Outcomes (GTO) is used to strengthens the knowledge, attitudes, and skills practitioners need to carry out evidence based programs. In GTO, staff receive ongoing technical assistance using the GTO implementation platform.
  Interventions: Other: Getting To Outcomes; Behavioral: Maintaining Independence and Sobriety Through Systems Integration, Outreach, and Networking (Veterans Edition)
- Getting to Outcomes Veterans (Experimental): Getting To Outcomes (GTO) is used to strengthens the knowledge, attitudes, and skills practitioners need to carry out evidence based programs. In GTO, staff receive ongoing technical assistance using the GTO implementation platform, that guides staff while delivering MISSION to Veterans.
  Interventions: Other: Getting To Outcomes; Behavioral: Maintaining Independence and Sobriety Through Systems Integration, Outreach, and Networking (Veterans Edition)

INTERVENTIONS:
Behavioral: Maintaining Independence and Sobriety Through Systems Integration, Outreach, and Networking (Veterans Edition) — MISSION-Vet has been developed to target mental health, substance abuse and related issues facing homeless Veterans through assertive outreach, psychoeducation, and linkages to community-based resources
  Other Names: MISSION-Vet
  Arms: Implementation as Usual Case Management; Implementation as Usual Veterans
Other: Getting To Outcomes — GTO strengthens the knowledge, attitudes, and skills practitioners need to carry out evidence based programs. GTO consists of a series of steps practitioners should follow in order to obtain positive results and then provides them with the guidance necessary to complete those steps with quality. According to GTO, "carrying out" an evidence based program includes a series of steps corresponding to three general areas: (1) planning - e.g., developing goals and performance targets, ensuring staff are trained in the evidence based program; (2) implementation - e.g., monitoring program activities, maintaining adherence to an evidence based program model, supervision; and (3) self-evaluation - e.g., tracking patient outcomes, using data to improve program operations.
  Other Names: GTO
  Arms: Getting to Outcomes Case Management
Behavioral: Maintaining Independence and Sobriety Through Systems Integration, Outreach, and Networking (Veterans Edition) — MISSION-Vet has been developed to target mental health, substance abuse and related issues facing homeless Veterans through assertive outreach, psychoeducation, and linkages to community-based resources
  Other Names: MISSION-Vet
  Arms: Getting to Outcomes Case Management
Other: Getting To Outcomes — GTO strengthens the knowledge, attitudes, and skills practitioners need to carry out evidence based programs. GTO consists of a series of steps practitioners should follow in order to obtain positive results and then provides them with the guidance necessary to complete those steps with quality. According to GTO, "carrying out" an evidence based program includes a series of steps corresponding to three general areas: (1) planning - e.g., developing goals and performance targets, ensuring staff are trained in the evidence based program; (2) implementation - e.g., monitoring program activities, maintaining adherence to an evidence based program model, supervision; and (3) self-evaluation - e.g., tracking patient outcomes, using data to improve program operations.
  Other Names: GTO
  Arms: Getting to Outcomes Veterans
Behavioral: Maintaining Independence and Sobriety Through Systems Integration, Outreach, and Networking (Veterans Edition) — MISSION-Vet has been developed to target mental health, substance abuse and related issues facing homeless Veterans through assertive outreach, psychoeducation, and linkages to community-based resources
  Other Names: MISSION-Vet
  Arms: Getting to Outcomes Veterans

SUMMARY:
A major goal for the Department of Veterans Affairs is to end Veteran homelessness by 2015. The VA's largest homelessness initiative is the joint Departments of Housing and Urban Development (HUD) and Veterans Affairs (VA) Supportive Housing program (HUD-VASH), which has been expanded greatly over recent years via the allocation of 30,000 Housing First vouchers between 2008 and 2010 and increased funding to hire 1,000 new program case managers. However, recent expansion has resulted in a number of implementation challenges including delays in the distribution of housing vouchers and dropout among program participants (25% of those housed in HUD-VASH drop out within a year). Much of this dropout can be attributed to untreated issues facing many Veterans enrolled in HUD-VASH. The most common among these untreated issues are mental health and substance use disorders. The presence of these disorders is due in large part to the fact that much of HUD-VASH case management focuses on housing placement and maintenance, with limited attention to mental health, substance abuse, and other related psychosocial issues, which when left untreated, negatively impacts voucher distribution and housing stability. This project will test an implementation model-Getting To Outcomes (GTO)-designed to assist in the delivery of an intervention for Veterans with co-occurring mental health and substance use disorders (MISSION-Vet) in the HUD-VASH program. The proposed study will compare implementation of MISSION-Vet currently being planned through VA Office of Patient Care Services to an enhanced approach using the GTO model. Thus, this project can contribute to ending all Veteran homelessness by 2015, a pledge made by President Obama.

DETAILED DESCRIPTION:
This project tests an implementation platform-Getting To Outcomes (GTO)-designed to assist in the delivery of an evidence-based intervention for Veterans with co-occurring mental health and substance use disorders (MISSION-Vet) in the HUD-VASH program. This project will be a cluster randomized controlled trial that compares implementation of MISSION-Vet augmented by GTO to MISSION-Vet Implemented as Usual (IU) at three of the largest HUD-VASH programs in the country: VA Central Western Massachusetts Healthcare System (Northampton, MA), VA Capitol Health Care Network (Washington, D.C.), and VA Eastern Colorado Health Care System (Denver, CO). This project will randomly assign 150 HUD-VASH case managers and 1106 Veterans on their caseloads who have received HUD-VASH vouchers and case management services into these two groups on a 1-year rolling admission basis determined by when the Veteran receives a housing voucher. The control group will receive MISSION-Vet in addition to HUD-VASH case management services and the intervention group will receive the same as the control, however the HUD-VASH case manager will have access to GTO implementation support.

To compare case managers implementing MISSION-Vet augmented with GTO to HUD-VASH case managers using IU strategies on the following variables: (1) fidelity to the MISSION-Vet intervention; (2) proportion of time the Veteran is housed; (3) mental health, substance use, and functional outcomes among Veterans; and (4) factors key to the successful deployment of a new treatment as specified by the Reach, Effectiveness, Adoption, Implementation, & Maintenance (RE-AIM) model.

Data will be collected on fidelity to MISSION-Vet in both IU and GTO groups. Data will also be collected on all subjects' substance use, overall mental health functioning, engagement in substance abuse treatment services, the length of time housed, and community participation. The investigators will collect data from individuals at baseline and three time points for up to one year. The investigators' data analysis strategy will be to use a repeated-measures model to test for the significance of the treatment-by-time interaction while accounting for the clustered design of case manager within site.

This study intends to serve a dual function of comparing implementation of MISSION-Vet currently being planned through VA Office of Patient Care Services to an enhanced implementation approach using the GTO model. The proposed research will help to guide policy and practice actions to implement MISSION-Vet with fidelity and effectiveness to achieve maximum outcomes among homeless Veterans.

ELIGIBILITY:
Inclusion Criteria:

VA HUD-VASH case manager at the Northampton, Denver, and Washington D.C. HUD-VASH programs

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2012-10-29 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2016-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Smelson, PsyD, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA; Matthew J. Chinman, PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (4):
- United States (4):
  - VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado
  - VA Central Office - HSR&D, Washington, DC, Washington D.C., District of Columbia
  - Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts
  - VA Central Western Massachusetts Healthcare System, Leeds, MA, Leeds, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] O K, Kline A, Sawh L, Fisher W, Rodrigues S, Kane V, Kuhn J, Ellison ML, Smelson DA. Unemployment and Co-occurring Disorders Among Homeless Veterans. Journal of Dual Diagnosis. 2013 Mar 27; 9(2):134-138.
- [Result] Smelson DA, Kline A, Kuhn J, Rodrigues S, O'Connor K, Fisher W, Sawh L, Kane V. A wraparound treatment engagement intervention for homeless veterans with co-occurring disorders. Psychol Serv. 2013 May;10(2):161-7. doi: 10.1037/a0030948. Epub 2012 Dec 17. PMID 23244030
- [Result] McInnes DK, Sawh L, Petrakis BA, Rao S, Shimada SL, Eyrich-Garg KM, Gifford AL, Anaya HD, Smelson DA. The potential for health-related uses of mobile phones and internet with homeless veterans: results from a multisite survey. Telemed J E Health. 2014 Sep;20(9):801-9. doi: 10.1089/tmj.2013.0329. Epub 2014 Jul 21. PMID 25046280
- [Result] Smelson DA, Chinman M, McCarthy S, Hannah G, Sawh L, Glickman M. A cluster randomized Hybrid Type III trial testing an implementation support strategy to facilitate the use of an evidence-based practice in VA homeless programs. Implement Sci. 2015 May 28;10:79. doi: 10.1186/s13012-015-0267-4. PMID 26018048
- [Result] Chinman M, McCarthy S, Hannah G, Byrne TH, Smelson DA. Using Getting To Outcomes to facilitate the use of an evidence-based practice in VA homeless programs: a cluster-randomized trial of an implementation support strategy. Implement Sci. 2017 Mar 9;12(1):34. doi: 10.1186/s13012-017-0565-0. PMID 28279207
- [Result] Smelson DA, Chinman M, Hannah G, Byrne T, McCarthy S. An evidence-based co-occurring disorder intervention in VA homeless programs: outcomes from a hybrid III trial. BMC Health Serv Res. 2018 May 5;18(1):332. doi: 10.1186/s12913-018-3123-9. PMID 29728148

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All case managers were invited to participate and verbally consented before randomization into the IU or the GTO group. 10 refused to participate.
Groups:
- MISSION-Vet - IU Case Management: Maintaining Independence and Sobriety Through Systems Integration, Outreach, and Networking (Veterans Edition):MISSION-Vet has been developed to target mental health, substance abuse and related issues faced by homeless Veterans through assertive outreach, psychoeducation, and linkages to community-based resources.
  Implementation as Usual (IU) - standard training on the MISSION model via a 1.5 hour webinar
- MISSION-Vet IU Veterans: Maintaining Independence and Sobriety Through Systems Integration, Outreach, and Networking (Veterans Edition):MISSION-Vet has been developed to target mental health, substance abuse and related issues faced by homeless Veterans through assertive outreach, psychoeducation, and linkages to community-based resources.
  Implementation as Usual (IU) - staff receive standard training on the MISSION model via a 1.5 hour webinar and then deliver MISSION services to Veterans
- GTO Case Management: Getting To Outcomes (GTO) is used to strengthens the knowledge, attitudes, and skills practitioners need to carry out evidence based programs. In GTO, staff receive ongoing technical assistance using the GTO implementation platform.
- GTO MISSION Veterans: Getting To Outcomes (GTO) is used to strengthens the knowledge, attitudes, and skills practitioners need to carry out evidence based programs. In GTO, staff receive ongoing technical assistance using the GTO implementation platform, while delivering MISSION services to Veterans.
Period: Overall Study
Arm/Group | MISSION-Vet - IU Case Management | MISSION-Vet IU Veterans | GTO Case Management | GTO MISSION Veterans
Started | 22 | 87 | 47 | 81
Completed | 22 | 87 | 37 | 81
Not Completed | 0 | 0 | 10 | 0

BASELINE CHARACTERISTICS:
Population: Limited baseline characteristics were collected for the Veteran population who received case management. Only age was collected for Veterans. No baseline characteristics were collected on the staff population.
Groups:
- MISSION-Vet - IU Veterans: Maintaining Independence and Sobriety Through Systems Integration, Outreach, and Networking (Veterans Edition):MISSION-Vet has been developed to target mental health, substance abuse and related issues faced by homeless Veterans through assertive outreach, psychoeducation, and linkages to community-based resources.
  Implementation as Usual (IU) - staff receive standard training on the MISSION model via a 1.5 hour webinar and then deliver MISSION services to Veterans.
- Enhanced Implementation Approach GTO Case Management: Getting To Outcomes (GTO) is used to strengthens the knowledge, attitudes, and skills practitioners need to carry out evidence based programs. In GTO, staff receive ongoing technical assistance using the GTO implementation platform.
- GTO Veterans: Getting To Outcomes (GTO) is used to strengthens the knowledge, attitudes, and skills practitioners need to carry out evidence based programs. In GTO, staff receive ongoing technical assistance using the GTO implementation platform, while delivering MISSION services to Veterans
- Total: Total of all reporting groups
Arm/Group | MISSION-Vet - IU Case Management | MISSION-Vet - IU Veterans | Enhanced Implementation Approach GTO Case Management | GTO Veterans | Total
Number analyzed (Participants) | 22 | 87 | 37 | 81 | 227
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: No baseline characteristics were collected on the case management population.
  years
    number analyzed (Participants) | 0 | 87 | 0 | 81 | 168
    (all) |  | 49.7 (10.8) |  | 55.9 (9.5) | 52.8 (10.6)
Sex/Gender, Customized [Number; unit: participants]
  Unknown | 22 | 87 | 37 | 81 | 227

OUTCOME MEASURES:

1. Primary Outcome: MISSION Fidelity Index
Description: The fidelity index assesses the presence or absences of activities within MISSION-Vet - DRT, peer led sessions, self-guided exercises, referrals made, and/or delivery of the workbook, to each participating Veteran. We analyzed fidelity as the percent of adoption of MISSION-Vet. The threshold for fidelity to adopt MISSION-Vet is 1 contact between the case manager and each participating Veteran. There is no composite score, fidelity to MISSION-Vet is if the case manager conducted at least 1 session with a Veteran.This measure was embedded into the VA Electronic Medical Record System. The investigators will assess the impact GTO has in facilitating adoption and use with fidelity to the MISSION-Vet 12-month service delivery platform, in comparison to implementation as usual.
Time Frame: 12-months
Population: Clinician fidelity to MISSION-Vet using IU or GTO. Only assessed Staff population.
Measure: Number; unit: percentage of MISSION-Vet staff use
Arm/Group | MISSION-Vet - IU Case Management | MISSION-Vet IU Veterans | GTO Case Management | GTO Veterans
Number analyzed (Participants) | 22 | 0 | 37 | 0
percentage of MISSION-Vet staff use | 0 |  | 68 |

2. Post Hoc Outcome: Number of Services Provided by Case Managers and Peers to Veterans
Description: Services provided by Case Managers OR Peers was computed by a count of the number of contacts between case managers OR peers and Veterans. This computed a total of all Veteran contacts, which was the sum of face-to-face contacts with Veterans and contacts on behalf of Veterans (described as Veteran contacts) with other stakeholders (e.g. family, medical providers). Assessed on a monthly basis for 12 months following study enrollment. These measures were obtained from the standardized monthly and quarterly status reports completed by case managers, which were extracted from HOMES. We used a linear-mixed effects model to calculate a Least-Squares Mean for each group at the study's end-point holding all variables in the model (Veteran age, Veteran sex, presence of an SMI diagnosis, employment) constant at their mean value.
Time Frame: 12 months
Population: All MISSION-Vet IU Veterans and GTO Veterans were analyzed from HUD-VASH data monitoring system HOMES (Homeless Operations, Management and Evaluation).
Measure: Least Squares Mean (Standard Error); unit: Number of Service Contacts
Arm/Group | MISSION-Vet - IU Case Management | MISSION-Vet IU Veterans | GTO Case Management | GTO Veterans
Number analyzed (Participants) | 0 | 87 | 0 | 81
Number of Service Contacts |  | 3.466 (2.824) |  | 3.469 (3.051)
Statistical Analysis 1: Comparison: MISSION-Vet IU Veterans vs GTO Veterans; Compared changes in service intensity among Veterans served by case managers in the GTO group relative to the comparison group of Veterans, by fitting a series of mixed-effects regression models. Final mixed-effect models for all outcomes included fixed terms for group (GTO group vs. comparison), time, group x time interaction as well as control covariates; Test type: Superiority or Other; p = .04, Mixed Models Analysis

3. Post Hoc Outcome: Drug and Alcohol Dependence
Description: Examined monthly alcohol and drug use by Veterans. Assessed on a monthly basis for 12 months following study enrollment. These measures were obtained from the standardized monthly and quarterly status reports completed by case managers, which were extracted from HOMES.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Monthly Substance Use
Arm/Group | MISSION-Vet - IU Case Management | MISSION-Vet IU Veterans | GTO Case Management | GTO Veterans
Number analyzed (Participants) | 0 | 87 | 0 | 81
Monthly Substance Use
  Drug Use |  | 1.291 (0.62) |  | 1.786 (0.588)
  Alcohol Use |  | 1.668 (0.79) |  | 2.278 (0.752)
Statistical Analysis 1: Comparison: MISSION-Vet IU Veterans vs GTO Veterans; Compared changes in alcohol dependence among Veterans served by case managers in the GTO group relative to the comparison group of Veterans, by fitting a series of mixed-effects regression models. Final mixed-effect models for all outcomes included fixed terms for group (GTO group vs. comparison), time, group x time interaction as well as control covariates; Test type: Superiority or Other; p = .21, Mixed Models Analysis
Statistical Analysis 2: Comparison: MISSION-Vet IU Veterans vs GTO Veterans; Compared changes in drug dependence among Veterans served by case managers in the GTO group relative to the comparison group of Veterans, by fitting a series of mixed-effects regression models. Final mixed-effect models for all outcomes included fixed terms for group (GTO group vs. comparison), time, group x time interaction as well as control covariates; Test type: Superiority or Other; p = .07, Mixed Models Analysis

4. Post Hoc Outcome: Predicted Values of Veteran Inpatient Hospitalizations for Medical and Mental Health Conditions
Description: Number of inpatient hospitalization for medical and mental health conditions. Assessed on a monthly basis for 12 months following study enrollment. These measures were obtained from the standardized monthly and quarterly status reports completed by case managers, which were extracted from HOMES. A dichotomous measure of whether a veteran experienced an inpatient hospitalization for medical or mental health conditions , and not a count of number of hospitalizations. Specifically, we used a mixed-effects logistic regression model to calculate a predicted values (i.e. a Least-Squares Mean) for each group/arm at the study's end-point holding all variables in the model (Veteran age, Veteran sex, presence of an SMI diagnosis, employment) constant at their mean value. Predicted value reported in log-odds (logit) units.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Inpatient Hospitalization Log Odds Units
Arm/Group | MISSION-Vet - IU Case Management | MISSION-Vet IU Veterans | GTO Case Management | GTO Veterans
Number analyzed (Participants) | 0 | 87 | 0 | 81
Inpatient Hospitalization Log Odds Units
  Medical Inpatient Hospitalizations |  | -6.597 (1.903) |  | -6.555 (1.498)
  Mental Health Inpatient Hospitalizations |  | -5.311 (6.008) |  | -3.825 (5.802)
Statistical Analysis 1: Comparison: MISSION-Vet IU Veterans vs GTO Veterans; Compared mental health inpatient hospitalizations among Veterans served by case managers in the GTO group relative to the comparison group of Veterans, by fitting a series of mixed-effects regression models. Final mixed-effect models for all outcomes included fixed terms for group (GTO group vs. comparison), time, group x time interaction as well as control covariates; Test type: Superiority or Other; p = .14, Mixed Models Analysis
Statistical Analysis 2: Comparison: MISSION-Vet IU Veterans vs GTO Veterans; Compared medical inpatient hospitalizations among Veterans served by case managers in the GTO group relative to the comparison group of Veterans, by fitting a series of mixed-effects regression models. Final mixed-effect models for all outcomes included fixed terms for group (GTO group vs. comparison), time, group x time interaction as well as control covariates; Test type: Superiority or Other; p = .19, Mixed Models Analysis

5. Post Hoc Outcome: Predicted Values of Veteran Emergency Department Visits for Medical and Mental Health Concerns
Description: Number of emergency department visits for medical and for mental health. Assessed on a monthly basis for 12 months following study enrollment. These measures were obtained from the standardized monthly and quarterly status reports completed by case managers, which were extracted from HOMES. A dichotomous measure of whether a veteran experienced an emergency department visit for medical or mental health conditions , and not a count of number of emergency department visits. We used a mixed-effects logistic regression model to calculate a predicted values (i.e. a Least-Squares Mean) for each group/arm at the study's end-point holding all variables in the model (Veteran age, Veteran sex, presence of an SMI diagnosis, employment) constant at their mean value. Predicted value reported in log-odds (logit) units.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Log Odd Units of Emergency Dept. Visits
Arm/Group | MISSION-Vet - IU Case Management | MISSION-Vet IU Veterans | GTO Case Management | GTO Veterans
Number analyzed (Participants) | 0 | 87 | 0 | 81
Log Odd Units of Emergency Dept. Visits
  Medical Emergency Dept Visits |  | -4.663 (3.063) |  | -3.983 (2.923)
  Mental Health Emergency Dept Visits |  | -7.96 (2.312) |  | -6.792 (1.779)
Statistical Analysis 1: Comparison: MISSION-Vet IU Veterans vs GTO Veterans; Compared changes in mental health emergency department visits among Veterans served by case managers in the GTO group relative to the comparison group of Veterans, by fitting a series of mixed-effects regression models. Final mixed-effect models for all outcomes included fixed terms for group (GTO group vs. comparison), time, group x time interaction as well as control covariates; Test type: Superiority or Other; p = .24, Mixed Models Analysis

6. Post Hoc Outcome: Estimated Proportion of Veterans Without Negative Housing Exits
Description: We obtained information on negative housing exits from the HUD-VASH Exit form, which is available in HOMES and tracks the dates and reasons for all exits from the program. We measured whether and when a Veteran experienced a negative housing over the period from study enrollment (i.e. the first date of MISSION-Vet for those served by case managers in the GTO group and the date of the first MISSION-Vet session provided to any Veteran at the appropriate study site for this in the comparison group) until the end of the study observation period; the maximum follow-up time was 2.4 years, but only for HUD-VASH Exits. A negative exit was defined as an exit from HUD-VASH that occurred due to non-compliance with case management, eviction, Veteran dissatisfaction with housing, inability to locate Veteran and incarceration. Kaplan-Meier survival curves to calculate an estimate of the proportion of Veterans in each arm/group not experiencing a negative exit from housing at the study's endpoint.
Time Frame: 12 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Proportion of Veterans
Arm/Group | MISSION-Vet - IU Case Management | MISSION-Vet IU Veterans | GTO Case Management | GTO Veterans
Number analyzed (Participants) | 0 | 87 | 0 | 81
Proportion of Veterans |  | 0.808 [0.694 to 0.883] |  | 0.884 [0.737 to 0.952]
Statistical Analysis 1: Comparison: MISSION-Vet IU Veterans vs GTO Veterans; We used Kaplan-Meier survival curves to estimate the extent and timing of negative housing exits over time and Cox proportional hazards regression to assess the relationship between membership in the GTO group and risk of experiencing a negative housing exit, adjusting for a set of relevant covariates; Test type: Superiority or Other; p = .481, Regression, Cox

ADVERSE EVENTS:
Arm/Group | MISSION-Vet - IU Case Management | MISSION-Vet - IU Veterans | GTO Case Management | GTO Veterans
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/87 | 0/37 | 0/81
Other Adverse Events (participants affected / at risk) | 0/22 | 0/87 | 0/37 | 0/81

LIMITATIONS AND CAVEATS:
First peer specialists were not readily available to teams in the IU condition in two of the three sites. Second, HOMES data on case managers reports. Third, we believe the services documented underrepresented the actual amount of services delivered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes